CLINICAL TRIAL: NCT02272556
Title: Investigating the Role of Polyol Pathway in the Central Nervous System
Brief Title: Investigating the Role of the Polyol Pathway in the Central Nervous System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1408014461
Record Dates: First submitted 2014-10-20; First posted 2014-10-23 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Subjects with Type 2 Diabetes (Active Comparator): Type 2 DM subjects with HbA1C > 7.5% treated with metformin, sulfonylurea, insulin or combination
  Interventions: Other: Brain MRS during hyperglycemic clamp; Other: Analysis of Metabolites in cerebrospinal fluid
- Non-Diabetic Obese (Active Comparator): Age-matched, non-diabetic obese (BMI > 30 kg/m^3) individuals
  Interventions: Other: Brain MRS during hyperglycemic clamp; Other: Analysis of Metabolites in cerebrospinal fluid
- Lean, healthy control subjects (Active Comparator): Age-matched, lean, healthy control subjects (BMI < 25 kkg/m^3)
  Interventions: Other: Brain MRS during hyperglycemic clamp; Other: Analysis of Metabolites in cerebrospinal fluid

INTERVENTIONS:
Other: Brain MRS during hyperglycemic clamp — All patients will undergo brain MRS at baseline and following 2 and 4 hours of hyperglycemia using the clamp technique
Other: Analysis of Metabolites in cerebrospinal fluid — All patients will have the option to undergo a lumbar puncture for analysis of metabolites in cerebrospinal fluid

SUMMARY:
Patients will undergo magnetic resonance spectroscopy (MRS) scanning to noninvasively measure intracerebral and plasma metabolite levels at baseline and following 2 and 4 hours of hyperglycemia. Subjects will also undergo a lumbar puncture at a separate occasion to assess cerebrospinal fluid levels of metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM with HbA1C treated with metformin, sulfonylurea, insulin, or combination OR age-matched, non-diabetic obese (BMI > 30 kg/m^2) OR age-matched lean, healthy control subjects (BMI < 25 kg/m^2)
* Age 18-55
* BMI 18-45 kg/m^2

Exclusion Criteria:

* Creatinine > 1.5 mg/dL
* Hgb < 10 mg/dL
* ALT > 2.5 x ULN
* Untreated thyroid disease
* Uncontrolled Hypertension
* Known Neurological Disorders
* Untreated Psychiatric Disorders
* Malignancy
* Bleeding Disorders
* Smoking
* Current or recent steroid use in last 3 months
* Illicit drug use
* Pregnancy, actively seeking pregnancy, or breastfeeding
* Inability to enter MRI/MRS

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2015-02; Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

PRIMARY OUTCOMES:
Metabolite Measurements by MRS | 4 hours post hyperglycemia
  metabolite levels will be measured by MRS

SECONDARY OUTCOMES:
Hunger Ratings | 4 hours post hyperglycemia
  Hunger will be measured using a visual analog scale
Satiety Ratings | 4 hours post hyperglycemia
  Satiety will be measured using a visual analog scale
Cognitive State | 4 hours post hyperglycemia
  Participants will be asked to complete basic cognitive testing using the mini-mental status exam and the Montreal cognitive assessment

OTHER OUTCOMES:
Cerebrospinal fluid cell count | 2 weeks post MRS testing
  Metabolite levels will be measure in collected spinal fluid
protein levels | 2 weeks post MRS testing
  Metabolite levels will be measure in collected spinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sherwin, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States